CLINICAL TRIAL: NCT07206394
Title: A Feasibility Trial of ScarWork on Post-breast Surgery Pain Syndrome (PBSPS) in Early Stage Breast Cancer Patients.
Brief Title: Feasibility Trial of ScarWork for Post-breast Surgery Pain Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: University of West London (Other)
Responsible Party: Principal Investigator, John Hughes, Associate Professor/ Head of Research, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 352185
Record Dates: First submitted 2025-09-11; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; ScarWork; feasibility study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will employ a pragmatic mixed methods randomised parallel-group exploratory design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ScarWork plus standard care (Active Comparator): Participant received up to 5 ScarWork sessions alongside usual standard of care
  Interventions: Other: ScarWork therapy
- Standard care (No Intervention): Participants continue with their usual standard of care and symptom management without additional intervention.

INTERVENTIONS:
Other: ScarWork therapy — ScarWork is a manual therapy technique involving gentle, hands-on massage of scar tissue. It is designed to improve the mobility and integration of scar tissue, reduce discomfort, and support tissue healing. The approach is tailored to each individual, based on the characteristics of their scar and sensitivity of the surrounding tissue. It is commonly used with people recovering from surgery or radiotherapy to help address symptoms such as pain, tightness, numbness, or altered sensation. In this study, participants in the intervention group will receive up to five ScarWork sessions delivered by a trained therapist, in addition to standard care.
  Arms: ScarWork plus standard care

SUMMARY:
Breast cancer is the most common cancer in women in the United Kingdom (UK). Most women are treated with a combination of surgery and radiotherapy. While these treatments are effective, they can cause ongoing breast pain for some, which can last months or even years. This long-term pain can have a major impact on quality of life, yet it is often overlooked and not well managed in routine care.

One in three women may still experience breast pain three years after treatment. The pain can come from scarring, tissue damage, or nerve changes caused by surgery and radiotherapy. Treatments for this pain are limited. Many patients are advised the pain will subside on its own or are given basic painkillers, which sometimes have limited impact.

ScarWork is a light-touch manual therapy, developed in the United States and aims to improve the way scars feel and look, reduce pain and tightness, and support healing. Although it has been available in the United Kingdom since 2014, there is very little research into whether ScarWork helps people who experience pain after breast cancer treatment.

This small study is a first step to see whether ScarWork could be a useful treatment for people who have experience breast pain after surgery and/or radiotherapy. The researchers want to know:

* Can this therapy be delivered in an NHS setting?
* Do people find it helpful?
* Is it worth doing a larger trial in the future?

Participants will be randomly placed in one of two groups: one group will continue with usual care, and the other will receive up to five sessions of ScarWork in addition to usual care. Everyone in the study will be asked to complete short questionnaires about their pain and other symptoms, before and after treatment, and again one month later. Participants will also be invited to talk about their experiences in a short phone or online interview.

This research will help show whether ScarWork might be a useful option for people dealing with breast pain after treatment. It will also help researchers design a larger trial in the future to test ScarWork more fully.

DETAILED DESCRIPTION:
Background Breast cancer is the most common cancer among women in the United Kingdom (UK). Each year, around 57,000 women are diagnosed. Many are treated with a combination of breast-conserving surgery (also known as a lumpectomy) and radiotherapy. These treatments are highly effective but can result in significant trauma to the breast tissue and skin, leading to long-term pain for some individuals.

Although short-term pain after surgery and radiotherapy is expected, some people go on to experience persistent and sometimes worsening pain long after the area has healed. This condition, often referred to as Post-Breast Surgery Pain Syndrome (PBSPS), can interfere with day-to-day life, emotional wellbeing, and recovery. Research suggests that as many as 40% of women still experience breast pain up to three years after treatment.

Despite this, there are currently few treatment options specifically targeting PBSPS. Most patients are offered basic pain relief or reassured that the pain will eventually fade. Surveys show that while most breast cancer specialists recognize this pain as a common issue, less than half routinely offer specific treatment for it.

ScarWork is a manual light touch therapy technique developed by therapist Sharon Wheeler in the United States. It involves gentle, targeted touch of scar tissue with the goal of improving tissue mobility, reducing pain and discomfort, and supporting healing. ScarWork has been used in the United Kingdom since 2014, but very little scientific research has been done to evaluate how effective it is, particularly for people experiencing post-surgery breast pain.

A previous evaluation found that cancer survivors who received ScarWork reported less pain, improved scar appearance and sensation, and a general reduction in symptoms. However, these findings were based on an early-stage service evaluation rather than a formal clinical trial.

About this study This feasibility study is designed to explore whether ScarWork can help people with early-stage breast cancer who are living with breast pain following surgery and/or radiotherapy. It will also assess whether delivering ScarWork within an NHS setting is practical and acceptable for both patients and healthcare providers.

The study is based at University College London Hospitals (UCLH) and is the first of its kind to investigate the use of ScarWork specifically for PBSPS in people treated with breast surgery.

Study design

Participants in this study will be randomly assigned to one of two groups:

* Standard care only, or
* Standard care plus ScarWork therapy (up to five individualised ScarWork sessions)

The ScarWork treatment will be tailored to each participant's needs, in keeping with typical clinical practice. Outcome measures will be collected at the beginning of the study, after the final ScarWork session, and again four weeks after the treatment ends. This will help the research team assess both immediate and longer-term effects of the therapy.

Participants will complete questionnaires about their pain, scar-related symptoms, and general wellbeing. They will be able to complete these online, by post, or over the phone with a researcher. Those in the ScarWork group may also be invited to take part in a short interview to share their experiences of the treatment and the study process.

The findings will help researchers decide whether a larger, more detailed clinical trial is possible and worthwhile in the future.

Importance of study Pain after breast cancer treatment is common but under-recognised and under-treated. This study addresses an important gap in care by exploring a therapy that could provide relief to thousands of people living with post-treatment pain. By assessing ScarWork in a structured NHS setting, the study also helps build evidence for how complementary therapies can be integrated into cancer aftercare in a safe and measured way.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Early breast cancer patients who have had breast surgery with curative intent
* Radiotherapy completed ≥ 6 months previously
* In remission with no sign of active local disease
* Registering a score of ≥3 on perceived pain intensity or pain burden on a 10-point numerical rating scale (NRS)
* English speaking and able to communicate reasonably well
* Able to give informed consent
* Willing to attend for regular treatment at RLHIM

Exclusion Criteria:

* History of post-breast surgery wound complications
* History of breast surgery unrelated to breast cancer treatment
* History of previous ScarWork therapy
* Diagnosis of lymphoedema
* Severe co-morbidities or cognitive disability
* Receiving physiotherapy for post-breast surgery pain syndrome at the time of trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
BREAST-Q Breast Conserving Therapy Module V2.0 | Baseline (Week 0, before first session), Week 12 (at final ScarWork session; control group same time point), Week 16 (4 weeks post-final session; control group same time point).
  A validated patient-reported outcome measure designed to evaluate outcomes among women undergoing breast conserving therapy, with the two overarching domains of 1) health-related quality of life and 2) patient satisfaction. Scales can be used selectively as appropriate to the research. For this study, we will measure:
  1. Quality of life domains using:
     * Psychosocial Well-being scale comprises 10 items that ask about body image and a woman's confidence in social settings, as well as emotional health and self esteem.
     * Sexual Well-being scale comprises 6 items that ask about feelings of sexual attractiveness and confidence relating to breasts.
     * Physical Well-being
       * Chest scale comprises 9 items measuring problems in the breast area (tightness, pulling, tenderness, pain), activity limitations and sleep problems due to discomfort.
       * Adverse Effects of Radiation scale
  2. Satisfaction with Breasts

OTHER OUTCOMES:
The Numeric Rating Scale | Baseline (Week 0, before first session), Week 12 (at final ScarWork session; control group same time point), Week 16 (4 weeks post-final session; control group same time point).
  The Numeric Rating Scale (NRS), a widely used measure of pain intensity, provides a simple method for assessing pain across diverse clinical settings11. The NRS typically employs an 11-point scale, ranging from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable (severe)." Patients are asked to select the number that best corresponds to their current level of pain intensity. The NRS's straightforward format allows for easy comprehension and administration, making it suitable for use with a wide range of patients, including those with cognitive impairments or language barriers. Its sensitivity to changes in pain intensity makes it a valuable tool for tracking response to ScarWork therapy and monitoring changes in pain. Total questions asked: 1
Patient Scar Assessment Questionnaire (PSAQ) | Baseline (Week 0, before first session), Week 12 (at final ScarWork session; control group same time point), Week 16 (4 weeks post-final session; control group same time point).
  A validated patient-reported outcomes measure for scarring designed to allow patients to convey their opinion regarding linear scars and designed to evaluate the effect of any novel scar therapy.12 Comprising five subscales (Appearance, Symptoms, Consciousness, Satisfaction with Appearance, and Satisfaction with Symptoms) it is regarded as reliable and valid measure of the patient's perception of scarring. PSAQ will provide data specific to how women feel about their scar(s). Total questions asked: 39
Measure Yourself Medical Outcome Profile (MYMOP) | Baseline (Week 0, before first session), Week 12 (at final ScarWork session; control group same time point), Week 16 (4 weeks post-final session; control group same time point).
  A validated, patient-generated (individualised) outcome questionnaire that is problem-specific but includes general wellbeing. Practical, reliable and sensitive to change, it has been widely used in studies investigating both complementary and orthodox interventions. Brief and simple to administer as part of the patient consultation, MYMOP captures the symptoms (physical, emotional or social) that the patient finds troublesome and in this study is intended to capture data about wider issues of scarring on daily life. 13 MYMOP provides informative data about what symptoms the patient finds most troublesome and is a means of gathering valuable data about the patients' experience and priorities. In addition, it contains a question about medications taken, which may provide useful information about pain relief and reduction of analgesics.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital for Integrated Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant confidentiality, as the dataset includes sensitive health information related to scar treatment outcomes. Aggregate or de-identified data may be available on request.